CLINICAL TRIAL: NCT02411799
Title: Prospective Multi-Center Follow-up of Patients Undergoing Instrumented Thoracic and Lumbar Arthrodesis Supplemented by the Implanet Jazz SystemTM
Brief Title: Instrumented Thoracic and Lumbar Arthrodesis Supplemented by the Implanet Jazz SystemTMd
Status: Terminated | Type: Observational
Why Stopped: Principal investigator has left the university. Research has been discontinued prior to study completion; Registry study: no analysis
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, H Francis Farhadi, MD, PhD, Assistant Professor, Ohio State University
Other Study IDs: 2014H0433
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Spondylolisthesis; Spinal Stenosis; Proximal Joint Kyphosis (PJK)
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Establish a data repository of patients who have undergone thoracic and/or lumbar instrumented arthrodesis procedure supplemented by the Implanet Jazz System.

DETAILED DESCRIPTION:
The purpose of this study is to create a data repository of patients who have undergone spinal arthrodesis procedures supplemented with the Implanet Jazz System. This device is designed to provide a stable interface between spinal constructs and the rods; it can be secured around vertebral structures (such as the lamina, transverse or spinous processes) from T1 to L5 and is intended to provide temporary stabilization as a bone anchor during the development of a solid bony fusion.

Patients who are candidates for hybrid thoracolumbar fixation with the Implanet Jazz System during arthrodesis surgery will be asked to participate in this protocol. Clinical data will be collected as indicated at 6 weeks, as well as 3, 6, 12, 24, 36 48, and 60 months post surgery in the database. Data collected will include demographic and surgical information, physiological data, neurological assessments and patient reported outcomes. This comprehensive database will allow for gathering of relevant information for potential future research use.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for spinal arthrodesis surgery (thoracic and/or lumbar) supplemented by the Implanet Jazz System are eligible to participate in this study.

Exclusion Criteria:

* Patients under the age of 18 are excluded because the investigators do not routinely perform spinal arthrodesis surgery on these patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for hybrid thoracolumbar fixation with the Implanet Jazz System during arthrodesis surgery.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2015-04; Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who have undergone thoracic and/or lumbar instrumented arthrodesis procedures supplemented by the Implanet Jazz System. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: H. Francis Farhadi, M.D., PhD., Principal Investigator — Assistant Professor
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Viswanathan VK, Kukreja S, Minnema AJ, Farhadi HF. Prospective assessment of the safety and early outcomes of sublaminar band placement for the prevention of proximal junctional kyphosis. J Neurosurg Spine. 2018 May;28(5):520-531. doi: 10.3171/2017.8.SPINE17672. Epub 2018 Feb 9. PMID 29424677